CLINICAL TRIAL: NCT05642624
Title: The PK/PD of Deoxycholic Acid Amphotericin B in Invasive Fungal Infection Patients With Sepsis/Septic Shock
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Songqiao Liu, MD, Southeast University, China
Other Study IDs: 2018ZDSYLL066-P01
Record Dates: First submitted 2018-11-18; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-11

CONDITIONS: Fungal Infection
Keywords: Blood Concentration; Deoxycholic Acid Amphotericin B; Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — Amphotericin B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sepsis group: invasive fungal infection patients who were diagnosed sepsis accoreding to the sepsis 3.0 guidlines.
  Interventions: Drug: Deoxycholic acid amphotericin B
- septic shock group: invasive fungal infection patients who were diagnosed septic shock accoreding to the sepsis 3.0 guidlines.
  Interventions: Drug: Deoxycholic acid amphotericin B

INTERVENTIONS:
Drug: Deoxycholic acid amphotericin B — Starting with 1mg and increasing by 5-25mg daily until the maintenance dose is 50mg/d.
  Other Names: amphotericin B

SUMMARY:
To explore the PK/PD of deoxycholic amphotericin B in invasive fungal infection patients with sepsis/septic shock;To compare the PK/PD of deoxycholic amphotericin B in invasive fungal infection patients with sepsis and septic shock.

DETAILED DESCRIPTION:
This was a single-center study.Patients who were diagnosed with in invasive fungal infection receieved deoxycholic acid amphotericin B during the study period.The information was recored including the general condition, infection index, PK/PD index and drug-related side effects.

ELIGIBILITY:
Inclusion Criteria:

Patients age more than 18 years old; Meet the criteria of Sepsis 3.0; Admitted to ICU; Patients were suspected or diagnosis of IFI,doctors determined the use of deoxycholic acid amphotericin B.

Exclusion Criteria:

Serum creatinine≥221umol/L; Deoxycholic acid amphotericin B or amphotericin B liposome were used for the past 7 days; Patients being treated with rifampicin; Unable to tolerate treatment of deoxycholic acid amphotericin B; BMI<18.5 or >30; Tumors; Pregnancy; Estimated time of survival<24h; Patients who participated in other studies within 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Sepsis admitted to ICU of Zhongda hospital
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
Cmax/MIC | 14 days
  PK/PD of Deoxycholic Acid Amphotericin B

SECONDARY OUTCOMES:
AUC24h/MIC | 14 days
  Concentration of Deoxycholic Acid Amphotericin B

CONTACTS AND LOCATIONS:
Overall Officials: Huang Yingzi, PHD, Principal Investigator — Zhongda Hospital
Locations (2):
- China (2):
  - Zhongda Hospital, Southeast University, Nanjing, Jiangsu
  - Zhongda Hospital, Nanjing, Jiangsu